CLINICAL TRIAL: NCT06221254
Title: Israeli IBD Research Nucleus (IIRN) Consortium: COBMINDEX Goes Forward- A Smartphone Application for Added Psychological Wellbeing in Crohn's Disease
Brief Title: A Smartphone Application for Added Psychological Wellbeing in Crohn's Disease
Acronym: COBMINDEX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other); Ben-Gurion University of the Negev (Other)
Responsible Party: Principal Investigator, Dr Doron Schwartz, Senior Physician, Department of Gastroenterology and Hepatology, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOR-0351-22-CTIL; SCRC22051 (Other: Soroka Clinical Research Center); MOH_2023-04-30_012589 (Registry Identifier: Ministry of Health MyTrial); 2203-05901 (Other Grant/Funding Number: The Leona M. and Harry B. Helmsley Charitable Trust)
Record Dates: First submitted 2023-08-31; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Crohn Disease
Keywords: Crohn's Disease; Health related quality of life; Cognitive behavioral therapy; Mindfulness; Immune regulation; Healthcare cost
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: 200 CD patients divided into two equal groups: Intervention and control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention- COBMINDEX application (Experimental): The intervention in this arm is to learn during the first 3 months, cognitive, behavioral and mindfulness based stress reduction with daily exercise using a research dedicated application. Than, additional 9 months of practicing daily only with the application.
  Interventions: Behavioral: COBMINDEX digital application
- Control- COBMINDEX with Human therapist (Active Comparator): The intervention in this arm is to learn during the first 3 months, cognitive, behavioral and mindfulness based stress reduction with daily exercise with human therapist, and than practicing daily only with the application.
  Interventions: Behavioral: Human therapist (Control)

INTERVENTIONS:
Behavioral: COBMINDEX digital application — COBMINDEX is a Cognitive, behavioral and mindfulness-based stress reduction with daily self-exercise. The intervention comprises of 7 sessions in which stress reduction techniques are learned. In this arm the Patient learns techniques and practices using digital application.
  Arms: Intervention- COBMINDEX application
Behavioral: Human therapist (Control) — COBMINDEX is a Cognitive, behavioral and mindfulness-based stress reduction with daily self-exercise. The intervention comprises of 7 sessions in which stress reduction techniques are learned. In this arm the Patient learns techniques from a human therapist (the comperator for learning from the application) and practices using digital application.
  Arms: Control- COBMINDEX with Human therapist

SUMMARY:
Psychological intervention by COBMINDEX application to reduce psychological stress among CD patients, fatigue and pain and improve the patients' well being, quality-of-life and disease-coping skills, as well as improvement of the patients' immunological profile and intestinal microbiome.

DETAILED DESCRIPTION:
200 patients will be randomly divided into two groups - 100 patients will learn and practice COBMINDEX by a human therapist-social worker and 100 patients will learn and practice COBMINDEX by a digital therapist using the COBMINDEX application.

In the first 3-months there will be an assessment of patient progress following randomization to human therapist or digital therapist using the application for learning and practicing. During this period, the group of the human social-worker will have a limited access to the application dedicated for daily exercises and assessment.

In the following 9-month period, all patients will practice using the application, each group by it's permissions.

There will be daily assessment of stress, pain, fatigue, well-being and frequent assessments of patients' medical, psychological, and immunological status.

Throughout the trial, adverse events and concomitant medications will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate and signed informed consent
* Hebrew-speaking
* Age 18-75
* Proven diagnosis of Crohn's disease, at least 3 months post-diagnosis
* Stable medical treatment for the last 3 months
* Any Harvey Bradshaw Index score
* Ability to operate a smartphone and cellular application

Exclusion Criteria:

* Diagnosis of ulcerative colitis or unclassified inflammatory bowel disease
* Planned surgery for Crohn's disease
* Surgery for Crohn's disease (excluding drainage of perianal abscess) in the last 3 months
* Psychiatric disease (schizophrenia, major depression or bipolar disorder)
* Alcohol or drug dependency (stable medical use of cannabinoids will be allowed)
* Pregnancy or planned pregnancy during study period
* Clinically significant comorbidity
* Former participation in COBMINDEX trials

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of application as compared to human therapist. | 12 months
  Develop a smartphone application that will teach the patient COBMINDEX and to determine whether the application will be as effective as the psychological intervention delivered by the therapists.
  the primary end point is SIBDQ disease specific HRQOL. 10 questions each scale 1-7 with range 7-70. higher is better.

SECONDARY OUTCOMES:
Cost-effectiveness | 12 months
  To determine the cost-effectiveness of the intervention as provided by application versus therapists by prospective monitoring of direct and indirect healthcare costs. A cost-effectiveness analysis to assess the value for money of the application versus therapist interventions will be performed using primary data collected from patients in the study. These data include information of utilization of healthcare services reported by patients. The cost of each service will be based on the Israel Ministry of Health List Price for health services. We will calculate indirect costs of lost productivity based on patient responses to the WPAI questionnaire. For each patient we will calculate the quality-adjusted life-year (QALY) based on responses to the SF-12 questionnaires
Effects of intervention on microbiome | 12 months
  alpha + beta diversity
Psychological improvment | 12 months
  Psychological self-report questionnaires
  WPAI- Work Productivity and Activity Impairment. four types of scores:
  1. Absenteeism
  2. Presenteesism
  3. Work productivty loss
  4. Activity Impairment all presented in presentage 0-100. higher is worse.
Psychological improvment | 12 months
  Psychological self-report questionnaires
  SWLS -The 5-item scale 0-7 "satisfaction with life scale" range 0-35 higher is better.
Psychological improvment | 12 months
  Psychological self-report questionnaires
  FACIT-CD, FACIT Fatigue Scale 13-item measure 0-4. range 0-52 higher is worse.
Psychological improvment | 12 months
  Psychological self-report questionnaires
  Brief COPE- The Brief-COPE is a 28 item self-report questionnaire range 0-4 higher is worse.
Psychological improvment | 12 months
  Psychological self-report questionnaires
  . BSI- The Brief Symptom Inventory a 53-item self-report inventory in which participants rate the extent to which they have been bothered (0 ="not at all" to 4="extremely")
Psychological improvment | 12 months
  Psychological self-report questionnaires
  PSS-4, Perceived Stress Scale 4. 4-item 0-4 score. range 0-16 higher is worse.
Psychological improvment | 12 months
  Psychological self-report questionnaires
  FMI, Freiburg Mindfulness Inventory 14 items range 0-4 higher is better.
Psychological improvment | 12 months
  Psychological self-report questionnaires
  SUDS- Subjective Units of Distress Scale. range 0-100 higher is worse.
disease severity measurement | 12 months
  C Reactive Protein mg/dl 0- 100 normal range 0-0.5 higher means more inflammation.
disease severity measurement | 12 months
  calprotectin (microg/g) 0-8000 normal range 0-50 higher means more inflammation.
disease severity measurement | 12 months
  Harvey Bradshaw Index - Crohn's disease symptom score range 0-36. higher is worse.

CONTACTS AND LOCATIONS:
Overall Officials: Ruthie Bekore, MPH, Study Director — Soroka University Medical Center; Ganit Goren, PhD, Study Director — Ben-Gurion University of the Negev
Locations (4):
- Israel (4):
  - Soroka University Medical Center, Beersheba
  - Rambam Health Care Campus i, Haifa
  - Belinson Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan

IPD SHARING:
Plan to Share IPD: No